CLINICAL TRIAL: NCT02344420
Title: Study to Compare the Cardiac Resynchronization Therapy (CRT) Response Rate in a Heart Failure (HF) Population With an Equal Distribution of Men and Women
Brief Title: Clinical Investigation on Differences in the Magnitude of CRT Response in WOmen Versus MEN
Acronym: BIOWOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOTRONIK-CR017
Record Dates: First submitted 2014-12-19; First posted 2015-01-26 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): As it is not a randomize trial there is only one study arm. Described interventions as echocariography, six minute walk test, Quality of Life test or self assessment score should be done in all patients.
  Interventions: Procedure: Echocardiography; Behavioral: Minnesota Living Heart Failure Questionnaire (MLHF); Procedure: Six minute walk test; Behavioral: Self assessment score

INTERVENTIONS:
Procedure: Echocardiography — The devices used within the study are the legally marked CRT devices from BIOTRONIK. CRT-P and CRT-D. As this is a post market study, all devices have a CE label and are used within their intended use. There are no study specific limitations nor mandatory device settings for the study.
  Subjects will undergo a standard echo assessment at baseline, 6 and 12 month follow up visit in order to assess the baseline characteristics and the changes as response to resynchronization.
Behavioral: Minnesota Living Heart Failure Questionnaire (MLHF) — MLHF will be obtained at baseline, 6 and 12 month FU. The goal of this questionnaire is to measure the subjects perception of how their heart failure and treatment affect their life. Questions are focused on physical, socio-economic, and psychological impairments that persons with congestive heart failure frequently attribute to their condition.
Procedure: Six minute walk test — The test will be performed at baseline, 6 and 12 month FU. The purpose of the test is to determine how far a patient can walk in six minute and relate it with the heart failure.
Behavioral: Self assessment score — patient will complete a self assessment questionnaire at 2, 6 and 12 month FU for the calculation of the Packer Score at 12 month.

SUMMARY:
BIOWOMEN is a study designed to compare the Cardiac Resynchronization Therapy (CRT) response rate in a Heart Failure (HF) population with an equal distribution of men and women. Different clinical variables will be collected (QRSd, Left Bundle Brunch Block (LBBB), HF etiology…) and compared in order to demonstrate that women may respond even better than men.

DETAILED DESCRIPTION:
Prospective, non-randomized, international, open, multicenter study. Patients that comply with the inclusion and exclusion criteria will be implanted with a BIOTRONIK CRT system.

The primary objective is to study the magnitude of CRT response measured as function of increase in Left Ventricular Ejection Fraction (LVEF) in order to demonstrate a superior CRT response in women.

The Secondary main objectives are:

* To study changes in major clinical variables during a 12M FU period in men and women
* To study how Left Ventricular End Diastolic Volume (LVEDV) and Left Ventricular End Systolic Volume (LVESV) change in men and women with CRT response
* To study CRT responders and value if there are significant gender differences at baseline with regards of presence of inter/intra ventricular dyssynchrony, HF etiology (ischemic versus non-ischemic cardiomyopathy), QRS morphology (LBBB vs. RBBB) and QRSd
* Observational assessment of how key baseline clinical variables are related to the patient's CRT response, to create a possible "gender specific" response model.
* Study the relationship between QRSd (amount of dyssynchrony) and CRT response in men and women

There are no study specific requirements for the implantation procedure of the CRT device; implantation will be performed according to the routine hospital's practice.

In order to obtain an equal distribution of males and females in the study population enrolled by the site, all the inclusions should be performed consecutively (based on the normal hospital flow of CRT candidates), but the difference in the enrolment rate by gender should not exceed > 2 by site at any time during the enrolment phase.

The study flowchart consists of a baseline assessment, implantation/pre-hospital discharge, 2 month Follow Up (FU), 6 month FU, 12 month FU, and final study.

Special assessments as echocardiography (echo), 6 minute walk test and Quality of Life test (QOL) will be performed at baseline, after 6 months and at one year follow-up.

12-lead electrocardiogram (ECG) will only be performed at baseline. Device testing, (Serious) Adverse (Device) Events ((S)A(D)E), and changes in medication will be collected during all planned study FUs throughout the duration of the study. A device interrogation outside the scheduled study FU window needs to be reported as unscheduled FU.

The timing for scheduled FUs is at 2 month, 6 month and 12 month after implantation (and pre-hospital discharge) with a time window of ± 1 month.

All the echo images and ECGs will be saved and sent to the respective Core Labs.

The estimated sample size is 494 patients: 247 men and 247 women.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a "De Novo" implantation of a CRT device according to ESC Guidelines
* Understand the nature of the procedure
* Give written informed consent

Exclusion Criteria:

* CRT Device replacements
* CRT upgrades
* Permanent / Persistent Atrial Fibrillation
* Age< 18 years
* Pregnant and breastfeeding women
* Subjects with irreversible brain damage from pre existing cerebral disease
* Subjects with acutely de compensated heart failure
* NYHA Class IV Heart Failure
* Heart transplantation six months prior to the enrolment or expected within next 3 months.
* Cardiac surgery 3 months prior to the enrolment or planned within next 3 months.
* Have a life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) changes at 12 month Follow Up (FU) | Baseline, 6 and 12 month
  To study the magnitude of Cardiac Resynchronization Therapy (CRT) response in women measured as a function of improvement in LVEF at 12moth FU in order to demonstrate that CRT response in women is better than men.

SECONDARY OUTCOMES:
Left Ventricular End Diastolic Volume (LVEDV) | Baseline, 6 and 12 month
  Reverse left ventricular remodelling is a promising surrogate measure of outcome after CRT. Left ventricular diastolic volumes will be compared between men and women to see if there are differences.
Left Ventricular End Systolic Volume (LVESV) | Baseline, 6 and 12 month
  Reverse left ventricular remodelling is a promising surrogate measure of outcome after CRT. Left ventricular systolic volumes will be compared between men and women to see if there are differences.
NYHA class | Baseline, 6 and 12 month Follow Up
  Clinical variable collect to evaluate patients heart failure
Quality Of Life test (QOL score) | Baseline, 6 and 12 month Follow Up
  Test perform by the patient to measure the perception of how is the heart failure and it´s treatment affected in their daily routine.
Patient's global self-assessment score | 2, 6 and 12 month Follow Up
  Questionnaire perform by the patient to evaluate how is the heart failure.
6 minute walk test | Baseline, 6 and 12 month Follow Up
  Test perform by the patient to evaluate how is the heart failure.
12 lead electrocardiogram (ECG) | Baseline
  A standard 12-lead ECG at 25 mm speed obtained. QRS with will be measured to relate with CRT response.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose MS Sancho-Tello, Physician, Principal Investigator — Hospital Universitario La Fe de Valencia
Locations (1):
- Hospital Clínico Universitario La Fe, Valencia, Spain